CLINICAL TRIAL: NCT03876860
Title: An Enhanced Vaginal Dilator Model to Improve Patient Adherence and Reduce Radiation-Induced Vaginal Stenosis: a Randomized Control Trial
Brief Title: An Enhanced Vaginal Dilator to Reduce Radiation-Induced Vaginal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Margaret Liotta (Other)
Responsible Party: Sponsor-Investigator, Margaret Liotta, Assistant Professor, Loyola University
Organization: Loyola University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 211334
Record Dates: First submitted 2019-02-27; First posted 2019-03-15 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Endometrial Cancer; Cervical Cancer; Vaginal Stricture; Radiation Toxicity
Keywords: Vaginal dilator; Vaginal stenosis
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: Randomized control trial with two arms including control arm and experimental arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Dilator (Active Comparator): Participants in control arm (active comparator) will receive standard vaginal dilator with standard set of instructions for dilator use, including both verbal and written instructions. Recommended dilator use is three-times weekly for ten minutes
  Interventions: Device: Standard Dilator
- Silicone Dilator (Experimental): Participants in experimental arm will receive standard vaginal dilator with addition of silicone ring with standard set of instructions for dilator use, including both verbal and written instructions. Recommended dilator use is three-times weekly for ten minutes
  Interventions: Device: Silicone Dilator

INTERVENTIONS:
Device: Silicone Dilator — Addition of silicone band to standard vaginal dilator
  Arms: Silicone Dilator
Device: Standard Dilator — Standard vaginal dilator
  Arms: Standard Dilator

SUMMARY:
This is a randomized control trial aimed to decreased radiation-induced vaginal stenosis in patients with endometrial or cervical cancer treated with post-operative external beam radiation therapy with or without brachytherapy. The intervention is an enhanced vaginal dilator model, including a silicone band placed at the desired depth of dilator insertion. The new model will be compared against the traditional vaginal dilator model used as our institutional standard of care. We hypothesize the enhanced model will improve adherence, correct use and efficacy of vaginal dilator use.

DETAILED DESCRIPTION:
Pelvic radiotherapy and vaginal brachytherapy play an integral role in managing gynecological malignancies, including endometrial and cervical cancer. Radiation-induced vaginal stenosis is a well recognized complication of radiation therapy and can result in painful, inadequate pelvic exams and sexual dysfunction. Current recommendations to prevent and manage vaginal stenosis include regular use of vaginal dilators, with our institutional recommendation being three times weekly for 10 minutes. Compliance varies among studies but is generally perceived to be low. Limited literature exists regarding ways to improve adherence and correct use of vaginal dilators. The goal of this study is to enhance the standard vaginal dilator model to improve patient outcomes. Eligibility includes women with endometrial or cervical cancer treated with post-operative external beam radiation therapy with or without brachytherapy. Patients will be randomized to either the standard vaginal dilator or an enhanced model. The enhanced dilator model includes the addition of a silicone band placed at the desired depth of vaginal dilator insertion, aimed to aide in correct insertion length. The primary aim of the study is patient adherence to vaginal dilator use. Secondary aims include vaginal length, CTCAE v5.0 grading scale for vaginal stricture, sexual function, self-reported comfort with use, and discomfort during office pelvic exams. Outcomes will be obtained based on physician reporting and patient surveys. All analyses will be completed by a biostatistician in the Clinical Research Office using SAS version 9.4.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of endometrial or cervical cancer
* Undergoing external beam radiation therapy with or without brachytherapy
* English-speaking

Exclusion Criteria:

* History or current presence of fistula

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Participant Adherence | 12 months
  Number of participants who use the vaginal dilator at least three times per week

SECONDARY OUTCOMES:
Vaginal Length | 12 months
  Vaginal length (in centimeters) measured using a POP-Q wooden stick
Vaginal stenosis grading scale | 12 months
  The vaginal stenosis grading scale is an ordinal scale ranging from 0 (no vaginal stenosis) to 3 (severe vaginal stenosis) as defined by the Common Terminology Criteria for Adverse Events Version 5.0 - vaginal stricture.
Change in female sexual function | 12 months
  The female sexual function index (FSFI) is a measure of sexual functioning in women. Scores range from 2 to 36 with higher scores indicating greater functioning. The baseline FSFI score is subtracted from the 12-month follow-up FSFI score for each participant.
Discomfort with pelvic exams | 12 months
  Discomfort with pelvic exams is measured using a visual analog scale (VAS) ranging from 0 (no discomfort) to 10 (severe discomfort)
Discomfort with dilator use | 12 months
  Discomfort with use of the dilator is measured using a visual analog scale (VAS) ranging from 0 (no discomfort) to 10 (severe discomfort)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret R Liotta, DO, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers

REFERENCES:
- [Background] Brand AH, Bull CA, Cakir B. Vaginal stenosis in patients treated with radiotherapy for carcinoma of the cervix. Int J Gynecol Cancer. 2006 Jan-Feb;16(1):288-93. doi: 10.1111/j.1525-1438.2006.00348.x. PMID 16445647
- [Background] Brand AH, Do V, Stenlake A. Can an educational intervention improve compliance with vaginal dilator use in patients treated with radiation for a gynecological malignancy? Int J Gynecol Cancer. 2012 Jun;22(5):897-904. doi: 10.1097/IGC.0b013e31824d7243. PMID 22552831
- [Background] Bruner DW, Lanciano R, Keegan M, Corn B, Martin E, Hanks GE. Vaginal stenosis and sexual function following intracavitary radiation for the treatment of cervical and endometrial carcinoma. Int J Radiat Oncol Biol Phys. 1993 Nov 15;27(4):825-30. doi: 10.1016/0360-3016(93)90455-5. PMID 8244811
- [Background] Hanlon A, Small W Jr, Strauss J, Lin LL, Hanisch L, Huang L, Bai J, Wells J, Bruner DW. Dilator Use After Vaginal Brachytherapy for Endometrial Cancer: A Randomized Feasibility and Adherence Study. Cancer Nurs. 2018 May-Jun;41(3):200-209. doi: 10.1097/NCC.0000000000000500. PMID 28437283
- [Background] Harkenrider MM, Block AM, Alektiar KM, Gaffney DK, Jones E, Klopp A, Viswanathan AN, Small W Jr. American Brachytherapy Task Group Report: Adjuvant vaginal brachytherapy for early-stage endometrial cancer: A comprehensive review. Brachytherapy. 2017 Jan-Feb;16(1):95-108. doi: 10.1016/j.brachy.2016.04.005. Epub 2016 May 31. PMID 27260082
- [Background] Jeffries SA, Robinson JW, Craighead PS, Keats MR. An effective group psychoeducational intervention for improving compliance with vaginal dilation: a randomized controlled trial. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):404-11. doi: 10.1016/j.ijrobp.2005.12.009. Epub 2006 Mar 20. PMID 16542794
- [Background] Kirchheiner K, Nout RA, Lindegaard JC, Haie-Meder C, Mahantshetty U, Segedin B, Jurgenliemk-Schulz IM, Hoskin PJ, Rai B, Dorr W, Kirisits C, Bentzen SM, Potter R, Tanderup K; EMBRACE Collaborative Group. Dose-effect relationship and risk factors for vaginal stenosis after definitive radio(chemo)therapy with image-guided brachytherapy for locally advanced cervical cancer in the EMBRACE study. Radiother Oncol. 2016 Jan;118(1):160-6. doi: 10.1016/j.radonc.2015.12.025. Epub 2016 Jan 9. PMID 26780997
- [Background] Kirchheiner K, Fidarova E, Nout RA, Schmid MP, Sturdza A, Wiebe E, Kranz A, Polterauer S, Potter R, Dorr W. Radiation-induced morphological changes in the vagina. Strahlenther Onkol. 2012 Nov;188(11):1010-7. doi: 10.1007/s00066-012-0222-0. Epub 2012 Sep 29. PMID 23053157
- [Background] Law E, Kelvin JF, Thom B, Riedel E, Tom A, Carter J, Alektiar KM, Goodman KA. Prospective study of vaginal dilator use adherence and efficacy following radiotherapy. Radiother Oncol. 2015 Jul;116(1):149-55. doi: 10.1016/j.radonc.2015.06.018. Epub 2015 Jul 8. PMID 26164775
- [Background] Miles T, Johnson N. Vaginal dilator therapy for women receiving pelvic radiotherapy. Cochrane Database Syst Rev. 2014 Sep 8;2014(9):CD007291. doi: 10.1002/14651858.CD007291.pub3. PMID 25198150
- [Background] Morris L, Do V, Chard J, Brand AH. Radiation-induced vaginal stenosis: current perspectives. Int J Womens Health. 2017 May 2;9:273-279. doi: 10.2147/IJWH.S106796. eCollection 2017. PMID 28496367
- [Background] Park HS, Ratner ES, Lucarelli L, Polizzi S, Higgins SA, Damast S. Predictors of vaginal stenosis after intravaginal high-dose-rate brachytherapy for endometrial carcinoma. Brachytherapy. 2015 Jul-Aug;14(4):464-70. doi: 10.1016/j.brachy.2015.03.001. Epub 2015 Apr 14. PMID 25887343